CLINICAL TRIAL: NCT00656409
Title: Conjugate Pneumococcal Vaccine in Ataxia Telangiectasia (AT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Purpose: Basic Science
Other Study IDs: 04MI07
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Ataxia Telangiectasia (AT)
Keywords: Ataxia telangiectasia,; Conjugated pneumococcal,; Prevenar,; Immunogenicity ,; Vaccine
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Conjugated pneumococcal vaccine (Prevenar)
  Other Names: Prevenar

SUMMARY:
Ataxia Telangiectasia (AT) is an autosomal recessive inherited condition caused by mutations in the ATM gene1. Patients suffer from neuro-degenerative problems, usually commencing in the second year of life, and affecting predominantly the cerebellum. They also develop the characteristic superficial telangiectases. Between 60 and 80% of affected children are immunodeficient. This is associated with deficiency of immunoglobulin A (IgA ) 2, of IgG23 and of antibody responses to pneumococcal polysaccharides4. Patients suffer recurrent sino-pulmonary infections but a recent study suggests poor correlation between immune status and immunological parameters5. If uncontrolled, recurrent pulmonary infections can contribute to the development of chronic lung disease and bronchiectasis. Preventative management includes continuous prophylactic antibiotic treatment in some with the need for replacement immunoglobulin therapy in only a small proportion of cases. Antibiotics have been reasonably effective in this situation but the emergence of resistance amongst community acquired pneumococcal isolates is a cause for concern. Appropriate immunisation strategies may also have a role.

This study is designed to look at antibody responses in a one versus two dose regimen in a cohort of AT patients recruited through the AT Society a national charitable organisation involved in providing support to families with this condition and in fostering education and research in the field.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of AT

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of vaccine

SECONDARY OUTCOMES:
Incidence of adverse reactions to vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom